CLINICAL TRIAL: NCT07021443
Title: The Effect of GLP-1 Analogues on Liver Steatosis and Fibrosis in Diabetic and Obese Patients in a Clinical Setting
Acronym: GLP1_NAFLD
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: GLP1_NAFLD
Record Dates: First submitted 2023-05-09; First posted 2025-06-15 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: non-interventional — non-interventional

SUMMARY:
This study aims to measure the effect of GLP-1 analogues on non-alcoholic fatty liver disease in patients with diabetes and/or obesity in a clinical context. Previous studies showed a positive effect of this medication, but these studies always took place in highly controlled settings. The question is to what extent liver values evolve in a non-controlled context. The real effect and thus the clinical utility of GLP-1 analogues will be measured.

DETAILED DESCRIPTION:
This study aims to measure the effect of GLP-1 analogues on non-alcoholic fatty liver disease in patients with diabetes and/or obesity in a clinical context. Previous studies showed a positive effect of this medication, but these studies always took place in highly controlled settings. The question is to what extent liver values evolve in a non-controlled context. The real effect and thus the clinical utility of GLP-1 analogues will be measured.

Patients in whom a GLP-1 analogue is started (as it would be outside the context of this study) may be recruited. Patients in whom a GLP-1 analogue was started 12 months earlier are also eligible. Once they were screened on the inclusion and exclusion criteria and they took into account and signed the informed consent, they can be definitively included. Participants will be followed for 12 months. There are 2 contact points, the first on the start day and the second after 12 months. During this period, serum markers of liver injury, type 2 diabetes and dyslipidaemia are monitored. With these, additional scores for hepatic steatosis (NAFLD liver fat score) and fibrosis (FIB-4 index) are calculated. A fibroscan (or elastography) is also performed to monitor the evolution of hepatic steatosis and fibrosis. The evolution of data is statistically analysed and hereby compared with the starting points.

ELIGIBILITY:
Inclusion Criteria:

* The patient is older than 18 years old.
* The patient has obesity, defined as a BMI of 30 or higher; and/or the patient suffers from T2DM, defined as a twice measured sfG of 125 mg/dl or higher, or a sfG of 100 to 125 mg/dl and a twice measured oral glucose tolerance test (OGTT) with a serum glucose (sG) of 200 mg/dl, or higher after 2 hours, or a random sG of 200 mg/dl or higher in symptomatic patients.
* The patient suffers from NAFLD in any stage, except cirrhosis. This has to be objec-tively diagnosed by either a CAP fibroscan (cutoff: > 238 dB/m); or by the calculated NAFLD liver fat score (cutoff: > -0,64), at least one of which has to be positive.
* The patient is starting a GLP-1 analogue as treatment for T2DM or obesity as would be prescribed outside of this study; or the patient has started a GLP-1 analogue as treatment for T2DM or obesity as would be prescribed outside of this study 12 months prior.
* If the patient is part of the retro-prospective branch data collected 12 months prior include at least a (CAP) fibroscan, a blood sample (measuring AST, ALT, GGT, sfG, sfI, HbA1c, HDL, LDL, total cholesterol and platelets) and a physical examination (measuring blood pressure, waist circumference, weight and length).

Exclusion Criteria:

* The patient suffers from alcohol induced fatty liver disease. Macrocytic anemia; de-creased vitamin B12 and folic acid; increased GGT, bilirubin, ferritin, TG and AST/ALT ratio can be used as serum markers of alcohol abuse. Interpretation of these results will be the left to the patient's clinician and their clinical expertise. Alterna-tively a weekly alcohol consumption of 21 units for men and 14 units for women can be used as a cutoff.
* The patient suffers from drug induced liver steatosis. Drugs warranting exclusion include glucocorticoids, amiodarone, tamoxifen, methotrexate, valproate, tetracycline and chemotherapeutic agents.
* The patient suffers from any other chronic liver disease. These will be checked trough lab test results in the patients file.
* The patient has liver cirrhosis, defined as a fibroscan score of 14 kPa or more; or a FIB-4 index of > 2,67. Elastography
* The patient is pregnant at time of enrolment or at any time during the study.
* The patient refuses to agree to the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from consultations in the diabetes- and obesity clinic in UZ Brussel. All diabetic and/or obese patients with objectified NAFLD starting a GLP-1 analogue, or whom have started a GLP-1 analogue 12 months prior, will be considered as possible candidates. Inclu-sion is definite after it is established that patients comply to all inclusion- and exclusion criteria and they agree to the informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2025-05-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Group: Obese and/or diabetic patients with objectified NAFLD starting a GLP-1 analogue
Period: Overall Study
Arm/Group | Study Group
Started | 50
Completed | 48
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 48
Age, Continuous [Median (Full Range); unit: years] | 58 [33 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
prevalence [Number; unit: participants]
  prevalence of obesity in patients participating | 48
  prevalence of T2DM in patients participating | 48
  prevalence of liver steatosis in patients participating | 48
Use of statins at initiation of GLP1a [Count of Participants; unit: Participants]
  patients using statins | 38
  patients not using statins | 10
Indication of GLP1a [Count of Participants; unit: Participants]
  T2DM | 46
  Obesity | 2

OUTCOME MEASURES:

1. Primary Outcome: Serum Markers (sfG) to Follow the Evolution of Liver Damage
Description: This study aims to measure the effect of GLP-1 analogues on liver steatosis and fibrosis in diabetic and obese patients in a real-life clinical setting. Serum markers will be used to follow the evolution of liver damage.
Time Frame: From time of infomed consent till 1 year after signing informed consent.
Population: To better understand potential therapeutic effects in patients with more pronounced liver involvement, subjects presenting with liver enzymes levels above the ULN at baseline were analyzed separately also.
  no AST under ULN was available at month 12 (m12) for 3 patients. no ALT under ULN was available at m12 for 1 patients. no GGT under ULN was available at m12 for 2 patients. no ALT above ULN was available at m12 for 2 patients. no GGT above ULN was available at m12 for 1 patients.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Study Group
Number analyzed (Participants) | 48
U/L
  AST under ULN at month 0: number analyzed (Participants) | 41
  AST under ULN at month 0 | 22.59 (7.997)
  ALT under ULN at month 0: number analyzed (Participants) | 35
  ALT under ULN at month 0 | 28.51 (14.716)
  GGT under ULN at month 0: number analyzed (Participants) | 38
  GGT under ULN at month 0 | 38.59 (22.542)
  AST under ULN at month 12: number analyzed (Participants) | 38
  AST under ULN at month 12 | 21.34 (8.515)
  ALT under ULN at month 12: number analyzed (Participants) | 34
  ALT under ULN at month 12 | 27.58 (15.448)
  GGT under ULN at month 12: number analyzed (Participants) | 36
  GGT under ULN at month 12 | 36.68 (22.534)
  AST above ULN at month 0: number analyzed (Participants) | 7
  AST above ULN at month 0 | 37.86 (2.61)
  ALT above ULN at month 0: number analyzed (Participants) | 13
  ALT above ULN at month 0 | 45.54 (13.457)
  GGT above ULN at month 0: number analyzed (Participants) | 10
  GGT above ULN at month 0 | 71 (22.857)
  AST above ULN at month 12: number analyzed (Participants) | 7
  AST above ULN at month 12 | 29.43 (13.501)
  ALT above ULN at month 12: number analyzed (Participants) | 11
  ALT above ULN at month 12 | 38.45 (17.218)
  GGT above ULN at month 12: number analyzed (Participants) | 9
  GGT above ULN at month 12 | 63 (30.054)

2. Primary Outcome: Fatty Liver Index (FLI)
Description: This study aims to measure the effect of GLP-1 analogues on liver steatosis and fibrosis in diabetic and obese patients in a real-life clinical setting. Serum markers will be used to calculate the Fatty Liver Index to evaluate steatosis.
  The Fatty Liver Index (FLI) (calculated using TG, GGT, abdominal waist circumference and BMI) was employed to monitor the risk for steatosis. FLI: < 30 as low risk, 30 to < 60 as intermediate risk, and ≥ 60 as high risk for liver steatosis.
Time Frame: From time of signing the ICF till 1 year after given informed consent
Population: no FLI was available at month 12 for 11 patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Group
Number analyzed (Participants) | 39
units on a scale
  FLI at month 0 | 88.92 (10.31)
  FLI at month 12: number analyzed (Participants) | 28
  FLI at month 12 | 80.39 (15.3)

3. Primary Outcome: FIB-4 Index
Description: This study aims to measure the effect of GLP-1 analogues on liver steatosis and fibrosis in diabetic and obese patients in a real-life clinical setting. Serum markers will be used to calculate the FIB-4 index to evaluate fibrosis.
  The FIB-4 index is a non-invasive tool used to assess the likelihood of advanced liver fibrosis in individuals, particularly those with conditions like non-alcoholic fatty liver disease (NAFLD) or type 2 diabetes. It combines age, aspartate aminotransferase (AST), alanine aminotransferase (ALT), and platelet count to generate a score that helps categorize patients into low, intermediate, or high risk for significant liver scarring.
  FIB-4 index: < 1,3 for patients < 64 years or < 2 for those > 64 years as low risk (F0-1 = mild fibrosis); 1,3 - 2,67 (< 64 years) or 2 - 2,67 (> 64 years) as intermediate risk (F2-3 = moderate fibrosis); and > 2,67 as high risk for advanced fibrosis (F4 = severe fibrosis to cirrhosis).
Time Frame: From time of signing the ICF till 1 year after given informed consent
Population: no FIB-4 score was available for 4 patients at month 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Group
Number analyzed (Participants) | 41
units on a scale
  FIB-4 at month 0 | 1.17 (0.54)
  FIB-4 at month 12: number analyzed (Participants) | 37
  FIB-4 at month 12 | 1.09 (0.56)

4. Primary Outcome: Serum Markers (HbA1c) to Follow the Evolution of Liver Damage
Description: as for outcome 1
Time Frame: From time of infomed consent till 1 year after signing informed consent.
Population: no HbA1c was available for 3 patients at month 12.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Study Group
Number analyzed (Participants) | 48
percentage
  HbA1c at month 0 | 8.16 (0.996)
  HbA1c at month 12: number analyzed (Participants) | 45
  HbA1c at month 12 | 7.14 (1.18)

ADVERSE EVENTS:
Time Frame: adverse events were followed for 1 year after informed consent was given.
Description: This study was purely observational for the patients. Everything in the study was done as part of the standard of care, therefor only SAE's were followed up. However no SAE occurred during the study.
Arm/Group | Study Group
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2023-04-28): https://cdn.clinicaltrials.gov/large-docs/43/NCT07021443/Prot_000.pdf